CLINICAL TRIAL: NCT05085301
Title: Clinical Performance of RapiGEN BIOCREDIT Malaria Ag RDTs for Detection of Plasmodium Infections in Patients With Symptoms Suggestive of Malaria
Brief Title: RapiGEN BIOCREDIT Malaria Ag RDTs WHO Prequalification Study
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: University of Khartoum (Other); Eijkman Institute for Molecular Biology (Other)
Responsible Party: Sponsor
Other Study IDs: MA016 RapiGEN
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Malaria; Diagnoses Disease; RDT
MeSH Terms: conditions — Malaria | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rapid diagnostic test — The performance of three index tests and two comparator tests will be compared to reference tests and gold standard microscopy.
  Other Names: BIOCREDIT

SUMMARY:
Since their introduction in the late 90's, rapid diagnostic tests (RDTs) have markedly improved our ability to control malaria; yet they have inherent limitations which include low sensitivity in Plasmodium vivax detection and inability to detect hrp2/3 gene deleted Plasmodium falciparum parasites. In addition, the spread of P. falciparum parasites lacking hrp2 gene jeopardizes the long-term use of P. falciparum-specific HRP2-based RDTs.

A partnership between RapiGEN, FIND, and the Bill and Melinda Gates Foundation (BMGF) is addressing these limitations by developing five novel malaria RDTs with improved pLDH and HRP2 detection.

RapiGEN has also developed three novel malaria RDTs - BIOCREDIT Malaria Ag Pf/Pv (pLDH/pLDH), BIOCREDIT Malaria Ag Pf (pLDH/HRP2) and BIOCREDIT Malaria Ag Pf (pLDH) - to address these drawbacks. The BIOCREDIT Malaria Ag Pf/Pv (pLDH/pLDH) is a combo test that detects P. falciparum and P. vivax on a single device. BIOCREDIT Malaria Ag Pf (pLDH/HRP2) targets both PfLDH and HRP2 antigens in P. falciparum; and BIOCREDIT Malaria Ag Pf (pLDH) has improved detection of pLDH in P. falciparum.

In countries with circulation of hrp2/3 deleted P. falciparum malaria parasites or high P. vivax burden, these improved RDTs may be invaluable in malaria elimination.

This study is a prospective and retrospective evaluation of RapiGEN's BIOCREDIT Malaria Ag RDTs in malaria-endemic countries to assess their clinical performance for detection of malaria. The purpose of this study is to provide a high level outline of the study design and conduct to support the collation of a data package for WHO Pre-Qualification proposed study.

DETAILED DESCRIPTION:
Malaria continues to create a major health burden in the tropics especially in Africa. Introduction of Artemisinin-based combination therapy (ACT) has dramatically improved the outcomes of morbidity and mortality of malaria cases. Introduction of RDTs as well dramatically influenced cases detection hence treatment. The situation in Sudan is not different from the general picture in all Africa and witness great reduction of deaths from malaria since the introduction of ACT in 2005 (1). The national protocol depends now on Giemsa stained slides microcopy or certified RDTs for diagnosis and ACT as first and second line of treatment (2).

Recommendation by World Health Organization (WHO) on parasitological confirmation of malaria cases by microscopy or rapid diagnostic tests (RDTs) before treatment increased the use and availability of RDTs worldwide (3).

Rapid diagnostic tests, since their introduction in the late 90's, have dramatically improved our ability to control malaria. Most RDTs are based on histidine-rich protein 2 (PfHRP2) or lactate dehydrogenase (pLDH), which are present in Plasmodium falciparum only and all human-infecting Plasmodium species respectively (4). However, the gradual spread of hrp2/hrp3-deleted mutants in several endemic countries in South America, Asia and Africa exerts a substantial potential impact on the utility of HRP2-based RDTs for case management in these settings.

Plasmodium lactate dehydrogenase (pLDH), on the other hand, appears as a good alternative to HRP2 as it is an essential protein expressed by all human-infecting Plasmodium species; however, pLDH-based RDTs were shown to perform poorly at low parasitaemia, which is common among patients infected with P. vivax, P. malariae and P. ovale species as well as in asymptomatic infections. Therefore, it is less preferred in endemic-countries. In these settings, malaria microscopy holds its reign as the standard of reference thanks to its low direct cost and ability to detect, quantify, and differentiate malaria parasites. However, it is also labour-intensive, time-consuming and expertise-demanding.

With the aim of addressing these limitations, RapiGEN has developed novel malaria RDTs, in partnership with FIND and the Bill and Melinda Gates Foundation (BMGF). RapiGEN developed BIOCREDIT Malaria Ag Pf/Pv (pLDH/pLDH), BIOCREDIT Malaria Ag Pf (pLDH/HRP2) and BIOCREDIT Malaria Ag Pf.

These may provide added value compared to currently available malaria RDTs, especially in settings where current tests prove to be insufficient due to hrp2 deletion or high burden of P. vivax malaria.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5 years old or older
* Presenting at the study site with fever or a history of fever during the preceding 48 hours
* Freely agreeing to participate by providing informed consent (and assent, if applicable)

Exclusion Criteria:

* Presence of symptoms and signs of severe illness and/or central nervous system infections as defined by WHO guidelines

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptoms suggestive of malaria seeking clinical care in health facilities. All patients will be assessed for eligibility of enrollment and those who full filled the criteria will be recruited in the study after signing an informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 674 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Point estimates of BIOCREDIT Malaria Ag Pf | 2 months
  Point estimates of diagnostic accuracy characteristics (sensitivity, specificity, NPV, PPV) with 95% confidence intervals for BIOCREDIT Malaria Ag Pf (pLDH/HRP2) and BIOCREDIT Malaria Ag Pf (pLDH) using the reference test (nPCR) as standard of truth for the detection of P. falciparum infections in patients with symptoms suggestive of malaria
Point estimate of BIOCREDIT Malaria Ag Pf/Pv (pLDH/pLDH) | 2 months
  Point estimates of diagnostic accuracy characteristics (sensitivity, specificity, NPV, PPV) with 95% confidence intervals for BIOCREDIT Malaria Ag Pf/Pv (pLDH/pLDH) using the reference test as standard of truth for the detection of P. falciparum and P.vivax infections in patients with symptoms suggestive of malaria

SECONDARY OUTCOMES:
Point estimates of comparator tests | 2 months
  Point estimates of diagnostic accuracy characteristics (sensitivity, specificity, NPV, PPV) with 95% confidence intervals of comparator tests using the reference test as standard of truth for the detection of P. falciparum and, P.vivax infections in patients with symptoms suggestive of malaria
Frequencies of hrp2/3 gene deletions | 2 months
  Frequencies of P. falciparum infections containing HRP2 and/or HRP3 mutations and the impact of those on HRP2-based RDT diagnostic accuracy

CONTACTS AND LOCATIONS:
Locations (2):
- Eijkman Institute for Molecular Biology, Jakarta, Indonesia
- Institute of Endemic Diseases, Medical Campus, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: Undecided